CLINICAL TRIAL: NCT07000656
Title: Prospective Evaluation of Micturition Desire-Relaxation Training Device for Treating Lower Urinary Tract Dysfunction in Children: A Randomized Controlled Pilot Study
Brief Title: Micturition Desire-Relaxation Training Device for Lower Urinary Tract Dysfunction in Children
Acronym: ICCS，LUTD，PNE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MR-31-24-03
Record Dates: First submitted 2025-05-24; First posted 2025-06-03 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Daytime Urinary Incontinence; Urinary Frequency; Lower Urinary Tract Dysfunction; Primary Nocturnal Enuresis
MeSH Terms: conditions — Diurnal Enuresis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham Intervention Group (Sham Comparator): This arm will enroll pediatric participants diagnosed with PNE, daytime urinary incontinence, or urinary frequency disorder according to the ICCS diagnostic criteria. Participants will follow the same baseline assessment protocol and stratified randomization based on sex, age, and enuresis frequency. They will undergo sham Micturition Desire-Relaxation Training, during which the device will remain inactive throughout each session. Training sessions will last approximately 10 minutes and be performed 5 to 10 times daily for a total of 4 weeks. A fluid intake and voiding diary will be submitted at the end of the sham training period. Participants will continue with follow-up assessments at 3 and 6 months post-intervention to evaluate natural symptom progression and recurrence, without further training.
  Interventions: Device: Sham device
- Micturition Desire-Relaxation Training (Experimental): This study includes children diagnosed with PNE, daytime urinary incontinence, and urinary frequency disorder according to the ICCS diagnostic criteria. Participants in the intervention group will undergo Micturition Desire-Relaxation Training, with each session lasting approximately 10 minutes, performed 5 to 10 times per day over an 8-week period. Changes in clinical symptoms and any adverse events will be systematically documented at baseline, and at 1 and 2 months during the intervention, as well as at 3 and 6 months post-treatment. For participants who achieve complete remission, caregivers will be asked to maintain daily records of enuresis episodes at 3 and 6 months after treatment to monitor potential recurrence.
  Interventions: Device: Micturition Desire-Relaxation Training Device

INTERVENTIONS:
Device: Micturition Desire-Relaxation Training Device — The device was developed by Shanghai Children's Medical Center in collaboration with Shanghai University of Engineering Science. It plays relaxation videos through a VR device and monitors the subjects' brain waves in real time using electroencephalography to evaluate their relaxation levels. The relaxation material is adjusted accordingly, and urination is recorded after training. Urine is collected and analyzed with a flow meter, generating a diagnostic report.
  Arms: Micturition Desire-Relaxation Training
Device: Sham device — Participants diagnosed with nocturnal enuresis, daytime urinary incontinence, and urinary frequency will be screened at Shanghai Children's Medical Center, and eligible patients will be recruited. Participants will be randomly assigned to the sham training group, in which they will wear the device without powering it on for 10 minutes each session, 5-10 times a day, for 4 weeks.
  Arms: Sham Intervention Group

SUMMARY:
Urine storage and voiding are fundamental physiological processes. In clinical settings, many cases of lower urinary tract dysfunction (LUTD) are closely associated with abnormal conditioned reflexes formed in the central nervous system during the urine storage or voiding phases. Relaxation, as a core physiological and psychological state, has been shown to promote effective urine storage and facilitate smooth voiding. By repeatedly training individuals to establish a new conditioned reflex linking the sensation of urinary urgency with a state of relaxation, it may be possible to improve bladder storage capacity and voiding function. Based on this concept, the investigators have developed the world's first Micturition Desire-Relaxation Training Device (Chinese Patent No.: ZL 2020 1 0397789.4). This study aims to evaluate the clinical efficacy of this device in treating LUTD in children.

DETAILED DESCRIPTION:
This randomized controlled trial aims to evaluate the clinical efficacy of the Micturition Desire-Relaxation Training Device in managing LUTD in children over a six-month period. A stratified block randomization method will be used, matching participants based on sex, age, and enuresis frequency. Eligible participants will be stratified by sex and age, and then randomly assigned (1:1) to either the intervention group or the sham intervention group using a computer-generated sequence. This method ensures group balance regarding baseline characteristics and enuresis severity.

In the intervention group, baseline voiding diaries will be completed prior to initiating training. The first session will be supervised by trained medical personnel, during which participants and caregivers will receive standardized instruction in device usage and bladder relaxation techniques. Each session will last approximately 10 minutes and will be conducted 3-4 times during the initial instructional phase. The device will then be provided for home use at no cost. Caregivers will receive remote support from study physicians during the intervention period. Home-based training will include 5-10 sessions per day, each lasting 10 minutes. Daily records-including images of urine output, session duration, and any adverse events-will be uploaded to a secure cloud platform for physician review. The intervention will continue for 8 weeks. Monthly records of fluid intake and voiding behavior will be maintained throughout the study. Follow-up assessments, including voiding diaries and enuresis questionnaires, will be performed at 3 and 6 months post-intervention to assess recurrence and long-term outcomes.

The sham group will follow identical baseline and training schedules; however, the device will remain inactive during each session. After 4 weeks, participants in this group will submit fluid intake and voiding records.

Primary outcome measures include the enuresis improvement rate, frequency of daytime urinary incontinence, and total number of voiding episodes within 24 hours. Secondary outcomes will include: scores for the micturition desire-awakening function, timing of enuresis events, bedtime and wake time, standardized bladder capacity, bladder variability rate, behavioral responses during incontinence, psychological/behavioral characteristics, and enuresis recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis according to the ICCS criteria:

   For nocturnal enuresis:

   At least one episode of involuntary nighttime urination per month for more than 3 months.

   No abnormalities in routine urinalysis. No period of bedwetting-free days lasting more than 6 months, except for organic diseases.

   For daytime urinary incontinence:

   At least one episode of intermittent urinary leakage during wakefulness per month for more than 3 months.

   No anatomical or neurological causes of urinary incontinence.

   For urinary frequency:

   The child experiences only urinary frequency and urgency, occurring during the day and before sleep, with intervals ranging from a few minutes to 1 hour. Each urination involves a small volume, less than 50% of the estimated bladder capacity [EBC (mL) = 30 + (age × 30)], typically less than 30 mL, sometimes just a few drops, while total daily urine volume remains within normal limits. When the child is engaged in play or focused, the intervals between urination are extended, and urinary frequency symptoms disappear after falling asleep.
2. Age: 5 to 18 years (inclusive), regardless of gender.
3. Voluntary participation: The child and their guardian must voluntarily participate in the trial and sign the informed consent form.

Exclusion Criteria:

1. Exclude enuresis caused by urinary tract infections, pinworms, myelitis, spinal cord injuries, epilepsy, cerebral developmental disorders, diabetes, and other neurological, urinary, or endocrine diseases, as well as transient enuresis due to excessive activity, mental fatigue, or excessive fluid intake before bedtime.
2. Exclude conditions causing urinary frequency such as neurogenic bladder, urinary tract infections, urethral syndrome, hypercalciuria, or metabolic diseases.
3. Patients who have participated in or are currently participating in other clinical trials within the past month.
4. Patients deemed unsuitable for participation in the clinical trial by the investigator.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Enuresis improvement rate | From enrollment to the end of treatment at 6 months
  The enuresis improvement rate is the sum of the complete and partial response rates. No response: <50% reduction. Partial response: 50 to 99% reduction. Complete response: 100% reduction.
Daytime urinary incontinence frequency | From enrollment to the end of treatment at 6 months
  The frequency of daytime urinary incontinence will be recorded using a voiding diary, with caregivers documenting each episode of urine leakage during waking hours. The daily frequency will be categorized using a study-specific ordinal scoring system as follows:
  Score 0: No daytime incontinence Score 1: ≤1 episode/day Score 2: 2-3 episodes/day Score 3: ≥4 episodes/day Higher scores indicate more severe daytime urinary incontinence.
Total number of voiding episodes in 24 hours | From enrollment to the end of treatment at 6 months
  The total number of voiding episodes per 24 hours will be calculated using a 3-day bladder diary. This includes both daytime and nighttime voids.

SECONDARY OUTCOMES:
Grade scoring of the micturition desire - awakening function | From enrollment to the end of treatment at 6 months
  The micturition desire-awakening function will be assessed using a study-specific, investigator-defined scoring system based on average nocturnal awakening ability. Scores range from 1 to 5, with higher scores indicating poorer awakening response to bladder signals. The scoring criteria are as follows: Score 5: Remains asleep most of the time after urination.
  Score 4: Only awakens after completely wetting the bed. Score 3: Awakens only after urinating a significant amount and then goes to the toilet to void the remaining urine.
  Score 2: Awakens after urinating a small amount and then goes to the toilet to void the remaining urine.
  Score 1: Awakened by the urge to urinate, without wetting the bed.
Enuresis recurrence rate | From enrollment to the end of treatment at 6 months
  Recurrence is defined as the reappearance of enuresis in previously cured patients, occurring more than once per month.
Timing of nocturnal enuresis episodes | From enrollment to the end of treatment at 6 months
  The timing of nocturnal enuresis episodes will be recorded during the night. If multiple episodes occur, the time of the first episode will be used for analysis.
Child's bedtime and wake time | From enrollment to the end of treatment at 6 months
  The child's bedtime and wake-up time will be recorded daily throughout the intervention period.
Standardized bladder capacity | From enrollment to the end of treatment at 6 months
  Standardized bladder capacity = bladder capacity/body surface area. Compare the standardized mean bladder capacity as well as the maximum and minimum daytime/nighttime bladder capacity changes from baseline to 6 months.
  The term mean daytime bladder capacity refers to the average volume of voided urine measured on the frequency volume chart throughout a 24-hour cycle.
  The term maximum/minimum daytime bladder capacity refers to the largest/smallest volume of voided urine measured on the frequency volume chart during the day. It excludes the first morning void.
  The term maximum/minimum nighttime bladder capacity refers to the largest/smallest volume of voided urine measured on the frequency volume chart during the night. It includes the first morning void.
Bladder variability rate | From enrollment to the end of treatment at 6 months
  Bladder variability rate = (standard deviation / average bladder capacity) * 100% The average bladder capacity and standard deviation will be calculated based on each voided volume from the 3-day bladder diary to determine the variability rate.
Behavioral response during daytime urinary incontinence episodes | From enrollment to the end of treatment at 6 months
  Behaviors of the child during episodes of daytime incontinence will be recorded, such as whether the child is aware of the leakage, embarrassed, attempts to hide it, or seeks help.
Child's psychological and behavioral characteristics | Assessed every 3 months from enrollment to the end of treatment at 6 months
  The psychological and behavioral characteristics of the child will be assessed using the Strengths and Difficulties Questionnaire (SDQ). This standardized instrument evaluates five domains: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior.
  The SDQ comprises 25 items, each rated on a 3-point scale (0 = "Not True," 1 = "Somewhat True," 2 = "Certainly True"). Subscale scores (range: 0-10) are calculated for each of the five domains. The Total Difficulties Score (range: 0-40) is derived by summing the scores of the first four subscales, excluding prosocial behavior. Higher total difficulties scores indicate more severe psychological problems, whereas higher prosocial scores reflect better social behavior.
  Total and subscale scores will be used to track changes in psychological and behavioral functioning throughout the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Micturition Desire-Relaxation Training, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bergmann M, Corigliano T, Ataia I, Renella R, Simonetti GD, Bianchetti MG, von Vigier RO. Childhood extraordinary daytime urinary frequency-a case series and a systematic literature review. Pediatr Nephrol. 2009 Apr;24(4):789-95. doi: 10.1007/s00467-008-1082-9. Epub 2008 Dec 18. PMID 19093136
- [Background] Austin PF, Bauer SB, Bower W, Chase J, Franco I, Hoebeke P, Rittig S, Vande Walle J, von Gontard A, Wright A, Yang SS, Neveus T. The standardization of terminology of lower urinary tract function in children and adolescents: update report from the Standardization Committee of the International Children's Continence Society. J Urol. 2014 Jun;191(6):1863-1865.e13. doi: 10.1016/j.juro.2014.01.110. Epub 2014 Feb 4. PMID 24508614